CLINICAL TRIAL: NCT06088602
Title: The Effect of Cryoneurolysis for the Treatment of Acute Postoperative Pain Following Total Knee Arthroplasty in High Pain Responders - A Randomized, Participant- and Observer-masked, Sham-controlled Trial
Brief Title: Cryoneurolysis for Acute Postoperative Pain Following Total Knee Arthroplasty
Acronym: CRISPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Deichmann Springborg, Dr., Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CryoTKA
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Postoperative Pain
Keywords: Cryoanalgesia; Acute postoperative pain; Total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: The patients will be randomized to 2 groups with 22 in each.
  Sham cryo (sham-group): Postoperative sham cryoneurolysis of the lower extremity.
  Cryoneurolysis (cryo-group): Postoperative cryoneurolysis of the superficial genicular nerves, i.e., the infrapatellar branches of the saphenous nerve (ISN) and the anterior femoral cutaneous nerve (AFCN).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Anaesthesiologist performing intervention is unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryo-group (Experimental): Postoperative cryoneurolysis of the superficial genicular nerves, i.e., the infrapatellar branches of the saphenous nerve (ISN) and the anterior femoral cutaneous nerve (AFCN).
  Interventions: Procedure: Cryoneurolysis
- Sham-group (Sham Comparator): Postoperative sham cryoneurolysis of the lower extremity.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Cryoneurolysis — Local anesthesia is injected in the skin. The superficial genicular nerves, more specifically the ISN and the AFCN, are visualized. A nerve stimulator is used to verify the visualized nerves., 2-3 ml of ropivacaine 5 mg/ml is injected around the nerves. After 5-15 minutes the effect is evaluated by assessing pain in the surgical area and asking the patient whether there is a pain relief. Following this evaluation, cryoneurolysis (Cryo-S, Metrum Cryoflex, Blizne Laszczynskiego, Poland) is performed unilaterally along a treatment line, the location of which was guided by visualization and palpation of anatomic landmarks. The ISN treatment line is located along the line that connects a point located 5 cm medial to the lower pole of the patella and a point located 5 cm medial to the tibial tubercle. The AFCN treatment line is located at one-third the length of the distance from the center of the patella to the top of the femur, with a width equal to the width of the patella.
  Arms: Cryo-group
Procedure: Sham — The exact same procedure as in the cryo-group is performed, except that the nerves are not frozen with the cryoneurolysis apparatus. Sound effects from the machine are replicated to give the patient the same experience as in the active intervention group.
  Arms: Sham-group

SUMMARY:
Cryoneurolysis is a regional anaesthetic technique that works by freezing peripheral sensory nerves. This technique can potentially provide analgesia after total knee arthroplasty (TKA). However, the technique is expensive and comprehensive. Pain 24 hours after surgery is associated with high amounts of late acute pain. Therefore, the aim of the current study was to compare the effect of postoperative cryoanalgesia with a sham treatment on acute postoperative pain in TKA patients with moderate to severe pain on the first postoperative day. The cryoanalgesia treatment will be performed 24 hours after surgery. Afterward, the patients will be followed for 24 weeks to determine the level of pain among other outcomes.

DETAILED DESCRIPTION:
Background Total knee arthroplasty (TKA) is a frequently performed procedure and is expected to increase in numbers due to the aging population and growing obesity rates. Fast-track regimes with multimodal opioid-sparing analgesia have improved postoperative outcomes. However, a subset of patients still experiences unsatisfactory levels of postoperative pain in the weeks following surgery, potentially delaying mobilization and recovery as well as increasing the need for opioid analgesics. Current recommendations for pain management following TKA according to the Procedure Specific Postoperative Pain Management (PROSPECT) Working Group include paracetamol, nonsteroidal anti-inflammatory drugs (NSAIDs), glucocorticoids, local infiltration analgesia, and single shot adductor canal block (ACB). However, the role of ACBs for pain after TKA has been under extensive debate in recent years. While an ACB may provide some pain relief, the duration of pain control is usually less than 24 h and the effect on length of stay (LOS) and opioid consumption is questionable.

In the past decades, cryoneurolysis has been used to treat acute pain following herniorrhaphy, tonsillectomy, and thoracotomy via the surgical incision. The emergence of percutaneous cryoprobes and the use of ultra-sound guided techniques has allowed for an increase in potential applications. Recently, the use of cryoneurolysis has gained attention as a potential regional anesthetic technique for the treatment of knee pain. Cryoneurolysis works by freezing peripheral nerves with temperatures in the range of -20⁰C to -100⁰C, causing a Wallerian degeneration of nerve axons distal to the treatment site. This process involves loss of the relative continuity of the axon and its covering of myelin but with a preservation of the surrounding endo-, peri-, and epineurium, thus allowing normal axonal regeneration and remyelination. Axons regenerate at a rate of 1-2 mm/day. Thus, resulting in a nerve block that typically will resolve with full recovery within weeks to months depending on the site of treatment.

The effect of cryoneurolysis on knee pain has been documented in a few studies. A randomized, double-blind, sham-controlled trial found that cryoneurolysis reduced symptoms of knee osteoarthritis for up to 150 days. A retrospective chart-review of 100 patients undergoing TKA found that cryoneurolysis significantly lowered LOS, reduced opioid consumption until 12 weeks after surgery, and reduced pain at the 2- and 6-weeks follow-up. Another retrospective analysis in 267 patients undergoing TKA found a comparable reduction in opioid requirements, pain, and LOS in patients treated with cryoneurolysis compared with historic controls. A recent RCT comparing cryoneurolysis to standard of care in 124 patients undergoing TKA found that cryoneurolysis reduced opioid consumption at 72 h, 6 weeks and 12-week follow-ups.

Although these findings are promising, cryoneurolysis is expensive and comprehensive, and might not be relevant in all patients receiving multimodal analgesia with COX-2 inhibitors, paracetamol, local infiltration analgesia, and high-dose steroid in a fully implemented enhanced recovery program. Several risk factors have been associated with a high pain response including age, gender, preoperative pain, psychological profile, and quantitative sensory testing (QST). However, when including postoperative pain in the prediction of acute pain, movement-evoked pain 24 h postoperatively is the best predictor for pain the week following surgery.

Using postoperative pain 24 h after surgery as a predictor of a sustained high pain response, we hypothesized that postoperative cryoanalgesia compared to a local anesthesia (LA) block with sham cryo treatment would reduce pain in patients with moderate to severe pain following TKA 2-7 days after surgery.

Aim To compare the effect of postoperative cryoanalgesia with a sham treatment consisting of LA block only on postoperative pain in the first week after surgery in TKA patients with moderate to severe pain on the first postoperative day.

Study plan In the outpatient clinic, the screening procedure will be performed among patients planned for TKA by the surgeons. Patients will be asked by orthopedic staff whether they may be contacted regarding the research project. The research staff will then contact potential patients either in person or via telephone. The written study information will be explained - either at the outpatient clinic or via telephone by the investigator.

All patients receive both spoken and written information. Information is given in a separate closed room without interruptions. All patients are given the chance of an additional meeting with the chance of bringing a relative. All patients must give a signed informed consent on paper prior to inclusion to participate in the study. The patient will sign the consent form on day 1 after surgery.

Perioperative treatment The pre-, intra-, and postoperative treatment-course follows the local operating procedures and common clinical guidelines implemented at the Dept. of Orthopedic Surgery, Hvidovre Hospital.

Preoperative standard treatment Preoperatively, the patient is examined by a specialized arthroplasty surgeon, and a basic preoperative health examination is done, along with a specialized anesthesiologic assessment planning the anesthesia for the TKA operation.

On the morning of surgery the patient will be given:

Celebra 400 mg Paracetamol 1 g

Anesthesia All included patients will receive general anesthesia or a neuraxial blockade in the form of a spinal anesthesia administered at level L2-L4, by injecting 2-3 ml of hyperbaric bupivacaine 0.5%. If spinal anesthesia is performed, perioperative sedation with propofol or other sedatives is optional and done in agreement with the patient. According to local guidelines, dexamethasone 0.3 mg/kg or 1 mg/kg IV rounded up to nearest 10 mg will be administered prior to surgery to patients with a pain catastrophizing scale score ≤ 20 or > 20, respectively. A supplement of local infiltration analgesia is administered directly into the surrounding tissue of the knee at the end of surgery, according to local operating procedure.

Tranexamic acid is administered as 1 g preoperatively, 1 g 3 h postoperatively, and 1 g in the surgical ward according to local operating procedure to prevent bleeding.

Surgical procedure A medial parapatellar approach will be used. No tourniquet is used. Following insertion of the prosthesis, local infiltration analgesia (LIA) with 200 mL 0.2% Ropivacaine will be injected in the posterior capsule, periarticular tissues and subcutaneous tissue. Joint capsule, subcutis and skin are closed with standard 3-layer closure and a compression bandage is applied. No drains are used. All patient will be operated with cemented components and patella resurfacing.

Standard postoperative treatment

The postoperative multimodal analgesic regimen consists of:

Celebra 200 mg x 2, for 7 days. Paracetamol 1 g x 4, for 7 days. Morphine 10-20 mg or opioid equivalents administered only as rescue opioids.

Intervention The intervention will take place after the inclusion at 20-32 h after TKA surgery. The procedure will be performed at the Dept. of Anesthesiology.

Cryoneurolysis mechanism of action Cryoneurolysis will be performed on the superficial genicular nerves (Cryo-S, Metrum Cryoflex, Blizne Laszczynskiego, Poland). The cryoprobe works by passing carbon dioxide at a relatively high pressure down the shaft, through a small orifice and into a closed tip at a much lower pressure. According to the Joule-Thomson effect, this drop in pressure causes a dramatic decrease in temperature which leads to a rapid expansion and absorption of heat. Afterwards the gas moves back up through a larger diameter tube. Importantly, this closed loop allows no gas to escape into the surrounding tissue. The intense cold created (approximately -70⁰C) causes a Wallerian degeneration, thereby reversibly destroying the nerve axon with retention of the endo-, peri-, and epineurium. Since the architecture of the nerve remains intact, the nerve axon can grow out along its normal path which occurs with approximately 1-2 mm/day. The drop in temperature cannot be lower than the boiling point for the gas used, which for carbon dioxide is -79⁰C. Irreversible degeneration of nerve tissue occurs at about -100⁰C which allows for a wide safety margin.

Procedure technique

Cryo-group:

The patient is placed in a supine position with a sheet between the upper and lower part of the body, thus blinding the patient from the intervention allocation. The procedure is performed using a linear array ultrasound probe. Local anesthesia is injected in the skin. The superficial genicular nerves, more specifically the ISN and the AFCN, are visualized. A nerve stimulator (Stimuplex HNS 12, B Braun, Melsungen, Germany) is used to verify the visualized nerves., 2-3 ml of ropivacaine 5 mg/ml is injected around the nerves. After 5-15 minutes the effect is evaluated by assessing pain in the surgical area and asking the patient whether there is a pain relief. Following this evaluation, cryoneurolysis (Cryo-S, Metrum Cryoflex, Blizne Laszczynskiego, Poland) is performed unilaterally along a treatment line, the location of which was guided by visualization and palpation of anatomic landmarks. The ISN treatment line is located along the line that connects a point located 5 cm medial to the lower pole of the patella and a point located 5 cm medial to the tibial tubercle. The AFCN treatment line is located at one-third the length of the distance from the center of the patella to the top of the femur, with a width equal to the width of the patella.

Sham-group:

The exact same procedure as in the cryo-group is performed, except that the nerves are not frozen with the cryoneurolysis apparatus. Sound effects from the machine are replicated to give the patient the same experience as in the active intervention group.

Study specific assessments Pain is rated by the patient before the intervention, after the initial LA injection, at home on days 2-7 and at the 2-, 4-, 12-, and 24 weeks follow-up via telephone.

A Visual Analog Scale (VAS 0-100) is used. On days 1-7 patients mark their pain in the electronic CRF twice a day (Appendix 5). If the patient is not able to complete the ratings electronically, a physical pain diary will be provided. Pain is rated by the patient at rest, during a 5-meter walk test, and during sleep. At the hospital and at the follow-ups patients are asked to rate their pain at rest and during a 5-meter walk test.

Use of rescue-analgesics (opioids) or other specific pain-relieving actions that differ from standard treatment is noted in the CRF.

The presence of dysesthesia or other side effects will be evaluated at each follow-up.

Other clinical data collected

* Demographical data (gender, age, height, weight, co-morbidity, American Society of Anesthesiologist (ASA) score)
* Preoperative opioids/strong analgesics
* Pain Catastrophizing Scale (PCS)
* Surgical data (date of surgery, indication, surgical time, procedure information, intraoperative bleeding, transfusion data, perioperative analgesics)
* Type and dosage of analgesics.
* Deviations from standard treatment
* Quality of sleep, lethargy, dizziness, and nausea, pre- and postoperative registration, on a NRS (0-10)
* Adverse events throughout the hospitalization and at each follow-up
* Neuropathic Pain Scale for Postsurgical Patients (NeuPPS)

Data protection The study will be conducted according to the General Data Protection Regulation and The Data Protection Act. All information will be treated confidentially, and all data will be pseudonymized with a code.

All research personnel are subject to professional secrecy. The investigators will keep an ID-list on all patients included in the study, containing full name, social security number and participant-ID.

A screening log is kept electronically in REDCap containing date of screening/surgery, age, reasons for not including in study on all patients screened for participation.

Collected data will be entered in the electronic CRF. This CRF and the EPJ will be made available for third parties in accordance with Danish Law. This means available for inspection by the Danish Medical Agency or other health authorities.

Patients will be informed that results will be stored and analyzed, and that anonymity will be respected. Data will always be stored in accordance with the regulations by DPA. Furthermore, participants will be informed of the possibility of inspection of the data from public authorities. Investigator ensures that the study follows the principles of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Primary unilateral total knee arthroplasty
* Ability to participate in the study (understand written and spoken Danish language, self-reported pain and satisfaction)
* Signed written informed consent form
* Pain (VAS 0-100 mm) ≥ 45 during a 5-meter walk test at 24 h (20-28h) postoperatively

Exclusion Criteria:

* Ongoing treatment of systemic glucocorticoids or other immunosuppressant treatment apart from inhaled steroids
* Insulin-dependent diabetes
* Pregnancy or breastfeeding
* Mental disability that could impair a patient's decision-making capability of giving informed consent and not enabling valid data collection.
* Patients with known diagnoses of schizophrenia, ongoing psychosis, bipolar disease and/or a history of ongoing anti-psychotic treatment.
* Patients with modulated pain-reception (experience) based on other diseases or injuries, e.g. spinal cord or brain injury, severe polyneuropathies or neurologic disorders.
* Posttraumatic osteoarthritis as reason for total knee arthroplasty
* Bleeding disorder
* Localized infection in the treatment area
* Cryoglobulinemia, cold urticaria, paroxysmal cold haemoglobinuria, or Raynaud's syndrome
* Perioperative peripheral nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Cumulated pain during walking days 2-7 | Days 2-7 after surgery
  Cumulated pain (VAS 0-100 mm) upon ambulation in a 5-meter walk test on days 2-7 postoperatively after surgery.

SECONDARY OUTCOMES:
Pain at follow-ups | 2-24 weeks after surgery
  Pain (VAS 0-100) during rest and during 5-meter walk test at the 2 weeks, 4 weeks, 12 weeks, and 24 weeks follow-up
Pain relief after block | 24 hours after surgery
  Pain relief immediately following blockade evaluated as ΔVAS 0-100 during a 5-meter walk test before and after the blockade
Cumulated pain during rest and night days 2-7 | Days 2-7 after surgery
  Cumulated pain at rest and during night from days 2-7
Quality of sleep | Days 2-7 after surgery
  Quality of sleep assessed by the patient on a scale of 0-10 from postoperative days 2-7
Dizziness | Days 2-7 after surgery
  Dizziness assessed by the patient on a scale of 0-10 from postoperative days 2-7
Fatigue | Days 2-7 after surgery
  Fatigue assessed by the patient on a scale of 0-10 from postoperative days 2-7
Nausea | Days 2-7 after surgery
  Nausea assessed by the patient on a scale of 0-10 from postoperative days 2-7
Use of rescue analgesics | 2 days to 24 weeks efter surgery
  Cumulative use of rescue-analgesics from days 2-7, and at 2 weeks, 4 weeks, 12 weeks, and 24 weeks follow-up
Oxford knee score | 12 weeks after surgery
  Oxford knee score at 12 weeks
Length of stay in hospital | Up to 24 weeks
  Length of stay in hospital, and reasons for prolonged stay (>1 postoperative day) registered as "Why still in hospital"
Reasons for re-admissions | 12 weeks
  Reasons for re-admissions within 12 weeks
Morbidity | 24 weeks after surgery
  Morbidity assessed as new illnesses or complications (4-, 12-, and 24 weeks follow-up by Electronic Patient Journal (EPJ) or telephone)
Mortality | 24 weeks after surgery
  Mortality (4-, 12-, and 24 weeks follow-up by Electronic Patient Journal (EPJ) or telephone)

CONTACTS AND LOCATIONS:
Overall Officials: Anders H Springborg, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data from all participants will be made available upon request after the study is published.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after the study is successfully published. There is no end date to the availability of the data.

REFERENCES:
- [Background] Husted H, Lunn TH, Troelsen A, Gaarn-Larsen L, Kristensen BB, Kehlet H. Why still in hospital after fast-track hip and knee arthroplasty? Acta Orthop. 2011 Dec;82(6):679-84. doi: 10.3109/17453674.2011.636682. Epub 2011 Nov 9. PMID 22066560
- [Background] Khan RS, Ahmed K, Blakeway E, Skapinakis P, Nihoyannopoulos L, Macleod K, Sevdalis N, Ashrafian H, Platt M, Darzi A, Athanasiou T. Catastrophizing: a predictive factor for postoperative pain. Am J Surg. 2011 Jan;201(1):122-31. doi: 10.1016/j.amjsurg.2010.02.007. Epub 2010 Sep 15. PMID 20832052
- [Background] Andersen LO, Gaarn-Larsen L, Kristensen BB, Husted H, Otte KS, Kehlet H. Subacute pain and function after fast-track hip and knee arthroplasty. Anaesthesia. 2009 May;64(5):508-13. doi: 10.1111/j.1365-2044.2008.05831.x. PMID 19413820
- [Background] Kehlet H, Joshi GP. The systematic review/meta-analysis epidemic: a tale of glucocorticoid therapy in total knee arthroplasty. Anaesthesia. 2020 Jul;75(7):856-860. doi: 10.1111/anae.14946. Epub 2019 Dec 4. No abstract available. PMID 31802486
- [Background] Callesen T, Bech K, Thorup J, Andersen J, Nielsen R, Roikjaer O, Kehlet H. Cryoanalgesia: effect on postherniorrhaphy pain. Anesth Analg. 1998 Oct;87(4):896-9. doi: 10.1097/00000539-199810000-00028. PMID 9768790
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Werner MU, Mjobo HN, Nielsen PR, Rudin A. Prediction of postoperative pain: a systematic review of predictive experimental pain studies. Anesthesiology. 2010 Jun;112(6):1494-502. doi: 10.1097/ALN.0b013e3181dcd5a0. PMID 20460988
- [Background] Barnard D. The effects of extreme cold on sensory nerves. Ann R Coll Surg Engl. 1980 May;62(3):180-7. PMID 7396346
- [Background] Mustola ST, Lempinen J, Saimanen E, Vilkko P. Efficacy of thoracic epidural analgesia with or without intercostal nerve cryoanalgesia for postthoracotomy pain. Ann Thorac Surg. 2011 Mar;91(3):869-73. doi: 10.1016/j.athoracsur.2010.11.014. PMID 21353017
- [Background] Urban JA, Dolesh K, Martin E. A Multimodal Pain Management Protocol Including Preoperative Cryoneurolysis for Total Knee Arthroplasty to Reduce Pain, Opioid Consumption, and Length of Stay. Arthroplast Today. 2021 Jul 12;10:87-92. doi: 10.1016/j.artd.2021.06.008. eCollection 2021 Aug. PMID 34286056
- [Background] Ilfeld BM, Gabriel RA, Trescot AM. Ultrasound-guided percutaneous cryoneurolysis for treatment of acute pain: could cryoanalgesia replace continuous peripheral nerve blocks? Br J Anaesth. 2017 Oct 1;119(4):703-706. doi: 10.1093/bja/aex142. No abstract available. PMID 29121277
- [Background] Joshi GP, Stewart J, Kehlet H. Critical appraisal of randomised trials assessing regional analgesic interventions for knee arthroplasty: implications for postoperative pain guidelines development. Br J Anaesth. 2022 Aug;129(2):142-144. doi: 10.1016/j.bja.2022.04.019. Epub 2022 May 24. PMID 35618537
- [Background] Lunn TH, Andersen LO, Kristensen BB, Husted H, Gaarn-Larsen L, Bandholm T, Ladelund S, Kehlet H. Effect of high-dose preoperative methylprednisolone on recovery after total hip arthroplasty: a randomized, double-blind, placebo-controlled trial. Br J Anaesth. 2013 Jan;110(1):66-73. doi: 10.1093/bja/aes345. Epub 2012 Sep 17. PMID 22986420
- [Background] Andersen KG, Christensen KB, Kehlet H, Bidstup PE. The Effect of Pain on Physical Functioning After Breast Cancer Treatment: Development and Validation of an Assessment Tool. Clin J Pain. 2015 Sep;31(9):794-802. doi: 10.1097/AJP.0000000000000156. PMID 25679946
- [Background] Riddle DL, Wade JB, Jiranek WA, Kong X. Preoperative pain catastrophizing predicts pain outcome after knee arthroplasty. Clin Orthop Relat Res. 2010 Mar;468(3):798-806. doi: 10.1007/s11999-009-0963-y. Epub 2009 Jul 8. PMID 19585177
- [Background] Rupp M, Lau E, Kurtz SM, Alt V. Projections of Primary TKA and THA in Germany From 2016 Through 2040. Clin Orthop Relat Res. 2020 Jul;478(7):1622-1633. doi: 10.1097/CORR.0000000000001214. PMID 32168057
- [Background] Cerantola Y, Valerio M, Persson B, Jichlinski P, Ljungqvist O, Hubner M, Kassouf W, Muller S, Baldini G, Carli F, Naesheimh T, Ytrebo L, Revhaug A, Lassen K, Knutsen T, Aarsether E, Wiklund P, Patel HR. Guidelines for perioperative care after radical cystectomy for bladder cancer: Enhanced Recovery After Surgery (ERAS((R))) society recommendations. Clin Nutr. 2013 Dec;32(6):879-87. doi: 10.1016/j.clnu.2013.09.014. Epub 2013 Oct 17. PMID 24189391
- [Background] Lavand'homme PM, Kehlet H, Rawal N, Joshi GP; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Pain management after total knee arthroplasty: PROcedure SPEcific Postoperative Pain ManagemenT recommendations. Eur J Anaesthesiol. 2022 Sep 1;39(9):743-757. doi: 10.1097/EJA.0000000000001691. Epub 2022 Jul 20. PMID 35852550
- [Background] Ju H, Feng Y, Yang BX, Wang J. Comparison of epidural analgesia and intercostal nerve cryoanalgesia for post-thoracotomy pain control. Eur J Pain. 2008 Apr;12(3):378-84. doi: 10.1016/j.ejpain.2007.07.011. Epub 2007 Sep 17. PMID 17870625
- [Background] Ilfeld BM, Preciado J, Trescot AM. Novel cryoneurolysis device for the treatment of sensory and motor peripheral nerves. Expert Rev Med Devices. 2016 Aug;13(8):713-25. doi: 10.1080/17434440.2016.1204229. Epub 2016 Jul 13. PMID 27333989
- [Background] Pabinger C, Lothaller H, Portner N, Geissler A. Projections of hip arthroplasty in OECD countries up to 2050. Hip Int. 2018 Sep;28(5):498-506. doi: 10.1177/1120700018757940. Epub 2018 May 21. PMID 29783896
- [Background] Romanini E, Decarolis F, Luzi I, Zanoli G, Venosa M, Laricchiuta P, Carrani E, Torre M. Total knee arthroplasty in Italy: reflections from the last fifteen years and projections for the next thirty. Int Orthop. 2019 Jan;43(1):133-138. doi: 10.1007/s00264-018-4165-7. Epub 2018 Oct 6. PMID 30293141
- [Background] Khanbhai M, Yap KH, Mohamed S, Dunning J. Is cryoanalgesia effective for post-thoracotomy pain? Interact Cardiovasc Thorac Surg. 2014 Feb;18(2):202-9. doi: 10.1093/icvts/ivt468. Epub 2013 Nov 11. PMID 24218494
- [Background] Mihalko WM, Kerkhof AL, Ford MC, Crockarell JR Jr, Harkess JW, Guyton JL. Cryoneurolysis before Total Knee Arthroplasty in Patients With Severe Osteoarthritis for Reduction of Postoperative Pain and Opioid Use in a Single-Center Randomized Controlled Trial. J Arthroplasty. 2021 May;36(5):1590-1598. doi: 10.1016/j.arth.2020.11.013. Epub 2020 Nov 14. PMID 33279353
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053
- [Background] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Background] Robinson SR, Purdie GL. Reducing post-tonsillectomy pain with cryoanalgesia: a randomized controlled trial. Laryngoscope. 2000 Jul;110(7):1128-31. doi: 10.1097/00005537-200007000-00011. PMID 10892682
- [Background] Erivan R, Villatte G, Dartus J, Reina N, Descamps S, Boisgard S. Progression and projection for hip surgery in France, 2008-2070: Epidemiologic study with trend and projection analysis. Orthop Traumatol Surg Res. 2019 Nov;105(7):1227-1235. doi: 10.1016/j.otsr.2019.07.021. Epub 2019 Oct 9. PMID 31606338
- [Background] Chan EY, Blyth FM, Nairn L, Fransen M. Acute postoperative pain following hospital discharge after total knee arthroplasty. Osteoarthritis Cartilage. 2013 Sep;21(9):1257-63. doi: 10.1016/j.joca.2013.06.011. PMID 23973139
- [Background] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Background] Paredes AC, Pinto JM, Almeida A, Pinto PR. Predictive value of quantitative sensory testing for acute and chronic postsurgical pain after total joint arthroplasty: a systematic review. Pain. 2022 Mar 1;163(3):e385-e400. doi: 10.1097/j.pain.0000000000002385. PMID 34224493
- [Background] Mejdahl MK, Christoffersens KB, Andersen KG. Development and Validation of a Screening Tool for Surgery-Specific Neuropathic Pain: Neuropathic Pain Scale for Postsurgical Patients. Pain Physician. 2019 Mar;22(2):E81-E90. PMID 30921980
- [Background] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT06088602/Prot_SAP_000.pdf